CLINICAL TRIAL: NCT07173855
Title: Effect of Protocolized Magnesium Replacement in Critically Ill Patients on Mortality and Atrial Fibrillation: the MAGNOLIA Randomized Controlled Trial
Brief Title: Effect of Protocolized Magnesium Replacement on Mortality and Atrial Fibrillation in Critically Ill Patients
Acronym: MAGNOLIA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Scarborough General Hospital (Other)
Collaborators: Scarborough Health Network (Unknown); Lakeridge Health Corporation (Other)
Responsible Party: Principal Investigator, Christopher Yarnell, Intensivist and Researcher, Scarborough General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICU-25-018
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-09

CONDITIONS: Critical Illness
Keywords: Critical illness; Magnesium; Atrial fibrillation; Protocols
MeSH Terms: conditions — Critical Illness; Atrial Fibrillation | interventions — Magnesium Oxide; alpha-glucoheptonic acid

STUDY DESIGN:
Intervention Model Description: Pragmatic comparative effectiveness trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lower target (>0.7mmol) (Other): Protocolized magnesium replacement according to magnesium level as follows: for 0.45 - 0.70mmol/L, magnesium sulfate 4g IV x 1 and repeat magnesium level the next day; for < 0.45mmol/L, magnesium sulfate 6g IV x 1, alert most responsible physician, and repeat level in 4 hours.
  Interventions: Drug: Magnesium sulfate administration
- Higher target (>0.95mmol/L) (Other): Protocolized magnesium replacement according to magnesium level as follows: for 0.75-0.95mmol/L, magnesium sulfate 2g IV x 1, magnesium oxide 420 mg po q12h x 2, or magnesium glucoheptonate 30mL po q12h x 2; for 0.45 - 0.74mmol/L, magnesium sulfate 4g IV x 1 and repeat magnesium level the next day; for < 0.45mmol/L, magnesium sulfate 6g IV x 1, alert most responsible physician, and repeat level in 4 hours.
  Interventions: Drug: Magnesium sulfate administration; Drug: Magnesium oxide; Drug: Magnesium glucoheptonate

INTERVENTIONS:
Drug: Magnesium sulfate administration — Magnesium sulfate is used in both arms for magnesium replacement.
Drug: Magnesium oxide — In the higher-target arm, magnesium oxide 420mg po q12h x 2 is one of the options available for magnesium replacement when magnesium levels lie between 0.75 and 0.95mmol/L.
  Arms: Higher target (>0.95mmol/L)
Drug: Magnesium glucoheptonate — Magnesium glucoheptonate 30mL po q12h x 2 is an oral option for magnesium replacement in the higher-target arm.
  Arms: Higher target (>0.95mmol/L)

SUMMARY:
In patients with critical illness, such as severe infections, heart attacks, or respiratory failure, most intensive care units (ICUs) measure magnesium levels and give supplemental doses of magnesium when levels are below certain targets. However, the best targets are unknown. The goal of this clinical trial is to study protocols for magnesium supplementation in people with critical illness, comparing a protocol with higher target level to a protocol with a lower target level.

The main question this study aims to answer is whether magnesium supplementation protocols targeting a higher or lower level lead to better 30-day survival and less atrial fibrillation.

Participants will not have to do any specific tasks, undergo any additional tests, or complete any surveys.

DETAILED DESCRIPTION:
Background: Measurement of serum magnesium levels, and administration of supplemental magnesium when levels are below target, is a common element of routine care for critically ill patients. However, targets for replacement vary, and the targets that lead to the best outcomes are unknown.

Methods: Multi-center open-label parallel group randomized controlled superiority trial of adult critically ill patients receiving protocolized magnesium replacement, comparing a higher target (>0.95mmol/L) to a lower target (>0.7mmol/L). The trial will be embedded into the electronic medical record (EMR) at 5 hospitals across 2 health networks in Ontario, Canada, with a shared EMR. Patients aged 16 years or older who have ICU admission orders and an order for the magnesium replacement protocol will be included. Patients with pre-eclampsia, sustained ventricular tachycardia, or neuromuscular junction disease will be excluded. The primary outcome will be an ordinal composite, evaluated at 30 days, composed of death and the number of days free of atrial fibrillation or flutter in ICU. Secondary outcomes will include ventricular arrhythmia and antiarrhythmics administered; receipt of vasopressors, ventilation, and new renal replacement therapy in ICU; lengths of ICU and hospital stay; hospital mortality at 60 and 90 days, magnesium levels, and magnesium supplementation. Analyses will use Bayesian regression with weakly skeptical priors and an intention-to-treat approach. Because both targets lie within the standard of care, the trial will use opt-out consent. Screening will be integrated with the EMR, such that when a patient meets inclusion criteria, a pop-up will appear for the ordering clinician. After the clinician confirms eligibility, the patient will be randomized and assigned to their target. Outcome ascertainment will occur within the EMR.

Discussion: This randomized controlled trial addresses an important uncertainty regarding routine care in the ICU with an EMR-embedded design. The innovative EMR-embedded design facilitates the large sample sizes and comprehensive, equitable recruitment needed for a trial evaluating a routine care intervention, and will lead to seamless integration with routine care upon trial completion.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years or older
* Admission orders written to a medical-surgical intensive care unit at a participating site
* Magnesium replacement protocol ordered

Exclusion Criteria:

* Prior enrollment in or withdrawal from MAGNOLIA trial
* Sustained ventricular tachycardia
* Pre-eclampsia
* Myasthenia gravis

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3253 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
30-day ordinal composite of hospital mortality and days free of atrial fibrillation in ICU | 30 days after enrollment.
  This is an ordinal outcome with 32 levels ranging from -1 (worst) to 30 (best). It is evaluated at 30 days. The worst outcome (-1) corresponds to mortality in hospital within 30 days from trial enrollment. Among patients who do not die in hospital by day 30, we count the number of days when they did not have atrial fibrillation in the ICU. For example, a survivor who never had atrial fibrillation in ICU would be scored as "30." A survivor who had 5 days of atrial fibrillation in ICU would be scored as "25." A patient who is discharged from hospital, either to home or transferred to another site, but is readmitted to a study hospital and dies within 30 days of enrollment, would be counted as having had hospital mortality. This stipulation is relevant because of the frequency of transfers between sites within a health network, due to regionalization of services such as vascular surgery, thoracic surgery, dialysis, and angiography.

SECONDARY OUTCOMES:
Organ-support free days | 30 days
  Number of days alive and free of invasive ventilation, vasopressors, and renal replacement therapy
ICU-free days | 30 days
  Number of days alive and not in ICU
Invasive ventilation-free days | 30 days
  Number of days alive and free of invasive ventilation
Vasopressor-free days | 30 days
  Days alive and not receiving vasopressors
Renal replacement therapy-free days | 30 days
  Days alive and not receiving renal replacement therapy in the ICU
Ventricular arrhythmia | 30 days
  Binary outcome noting the occurence of either sustained ventricular tachycardia or ventricular fibrillation in ICU (1), or not (0).
Intravenous antiarrhythmics | 30 days
  Binary variable noting administration of intravenous antiarrhythmics in ICU (1) or not (0). Intravenous antiarrhythmics include amiodarone, metoprolol, esmolol, diltiazem, procainamide, lidocaine, flecainide, adenosine, digoxin.
Magnesium and potassium levels in ICU | 30 days
  Daily levels of magnesium and potassium in ICU
Magnesium administrations | 30 days
  Magnesium administrations while in ICU (number per day)
Fluid balance | 30 days
  Daily fluid balance (sum of all liquid intakes minus the sum of all liquid outputs).
DOOR 1: Death and arrhythmia | 30 days
  This is a desirability of outcome ordinal ranking (DOOR) outcome. The possible binary levels are, from worst to best: death, ventricular arrhythmia, atrial fibrillation or flutter, none of the above.
DOOR 2: Survival, organ dysfunction, hospitalization, discharge | 30 days
  This is a desirability of outcome ordinal ranking (DOOR) outcome. The binary levels are, ordered from best to worst: discharge home, discharge to location other than home, ongoing hospital admission, persistent organ dysfunction in ICU, death.
Hospital mortality | 60 days
  Hospital mortality
Hospital mortality | 90 days
  Hospital mortality
Hospital length of stay | 90 days
  Length of hospitalization, including transfers within the health network.
Discharge destination | 90 days
  Categorical variable noting discharge destination on index hospitalization (eg home, retirement home, long-term care, acute care hospital, etc).
Magnesium administrations - by mass | 30 days
  Elemental magnesium administered (g per day)
Magnesium administrations - route | 30 days
  Route of magnesium administrations each day (PO vs IV)

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - Lakeridge Health Ajax-Pickering, Ajax, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Scarborough Centenary Hospital, Toronto, Ontario
  - Scarborough General Hospital, Toronto, Ontario
  - Scarborough Birchmount Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be posted in the Health Data Nexus (https://healthdatanexus.ai/) deidentified data repository overseen by the University of Toronto Temerty Centre for Artificial Intelligence Research and Education in Medicine. This will allow credentialed access to deidentified individual patient data.
Supporting Information: Study Protocol
Time Frame: Deidentified data will be posted in the Health Data Nexus repository after publication of the primary trial results.
Access Criteria: Credentialed access to the Health Data Nexus is available to anyone who fulfills the requirements, including an ethics course (TCPS2 2022) and signing a data use agreement.
URL: https://healthdatanexus.ai/